CLINICAL TRIAL: NCT02953418
Title: A Multicenter Trial of Endoscopic Radiofrequency Ablation for High-grade and Low-grade Intraepithelial Squamous Neoplasia Using the Barrx™ Flex Radiofrequency Ablation System
Brief Title: RFA for Flat Type High-grade and Medium-grade Intraepithelial Squamous Neoplasia
Acronym: REACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment taking longer than expected.
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVB3050540
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Squamous Cell Neoplasia (ESCN)
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Radiofrequency ablation (Experimental): Step-wise endoscopic RFA with the Barrx™ Flex Radiofrequency Ablation System using will be performed in 3 month intervals up to 12 months.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — RFA
  Other Names: The Barrx™ Flex Radiofrequency Ablation System

SUMMARY:
Multicenter, prospective cohort clinical trial in greater China

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-85 years of age
2. Patient has evidence of ESCN, within the last 3 months, patient demonstrated a new diagnosis or a reconfirmed diagnosis of squamous MGIN and/or HGIN of the esophagus
3. On endoscopic examination, subject has at least one USL that measures at least 3 cm in at least one dimension and greater than ¼ of the esophageal circumference and has MGIN or HGIN on biopsy, confirmed by central pathologist
4. All lesions in the esophagus are completely flat (Paris type 0-IIb), both on WLE and Lugol's chromoendoscopy
5. The maximum allowable linear length of "USL-bearing esophagus" is 12 cm
6. Baseline endoscopic ultrasound (EUS) (if applicable) shows no exclusionary findings for the trial
7. Computed Tomography )CT( scan of chest and upper third of the abdomen (if applicable) shows no exclusionary findings for the trial
8. Based on the judgment of the study endoscopist, the patient is eligible for treatment, follow-up endoscopy, and biopsy as required by the protocol
9. EMR or ESD occurred > 3 months before enrollment, patients may be eligible for the study if procedure was curative (negative margins and no risk of lymph node involvement) and the patient has no other findings concerning for cancer
10. The subject is willing to provide written, informed consent to participate in this clinical study and understands the responsibilities of trial participation

Exclusion Criteria:

1. Patient has esophageal squamous cell carcinoma (ESCC)
2. Any non-flat (Paris type 0-I, 0-IIa, 0-IIc, 0-III) abnormalities anywhere in the esophagus
3. Any abnormalities under WLE, Lugol's chromoendoscopy or NBI that are suspicious for ESCC anywhere in the esophagus (e.g. 'pink sign' USL, defined as a color change after Lugol's staining: initially whitish yellow and pink 2-3 minutes later)
4. Any USL with MGIN or worse on biopsy outside the treatment area
5. Esophageal stricture preventing passage of a therapeutic endoscope
6. Prior endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) which occurred < 3 months before enrollment
7. Any esophageal dilation in the past 12 months
8. Any history of a non-squamous cell cancer of the esophagus, or any history of a squamous cell cancer of the esophagus (any stage)
9. Any previous ablative therapy within the esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment, or other) or any radiation therapy to the esophagus
10. Previous esophageal surgery, except fundoplication without complications (i.e., no slippage, dysphagia, etc.)
11. Evidence of esophageal varices detected within last 6 months or at initial RFA procedure
12. Patient has active reflux esophagitis grade C or D
13. Evidence of eosinophilic esophagitis on endoscopy and/or histology
14. Inner diameter of the esophagus measuring <18 mm
15. Report of uncontrolled coagulopathy with international normalized ratio (INR) > 2 or platelet count <75,000 platelets per µL (note: a complete blood count is not required for all subjects in this study)
16. Patient is using anti-thrombotic agents that cannot be discontinued 7 days before and after therapeutic sessions
17. Patient has an implantable pacing device (examples: automated implantable cardioverter defibrillator, neurostimulator, cardiac pacemaker) and has not received clearance for enrollment in this study by specialist responsible for the pacing device
18. Patient has life expectancy less than 5 years
19. Patient suffers from psychiatric or other illness and/or has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post- treatment instructions, or follow-up guidelines
20. Patient is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity)
21. The subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
22. Patient is pregnant or has plans to become pregnant in the ensuing 12 months (confirmation of non-pregnant status in women of child-bearing age and ability required with urine or blood test to be eligible)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cafaro, RN, Study Director — Medtronic Gastrointestinal & Hepatology
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Ablation
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.41 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 34
Height (cm) [Mean (Standard Deviation); unit: cm] | 162.88 (7.79)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 64.93 (10.30)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Complete Response (CR)
Description: The primary endpoint is the percentage of subjects with "complete response (CR)", defined as complete eradication of squamous histological abnormalities (MGIN or worse) within the treatment area (TA) at 12 months after the initial treatment session
Time Frame: 12 month
Population: As the study was terminated early, only 8 subjects completed 12 month follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 8
Participants | 8

2. Secondary Outcome: Complete Response at Three Months
Description: Number of patients with a CR after primary RFA, defined as absence of MGIN or worse in any of the biopsies from the treatment area at the three months visit
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 34
Participants | 5

3. Secondary Outcome: Complete Response Within the Treatment Area
Description: Number of patients demonstrating complete response within the treatment area (TA), defined as detection of ESCC in biopsy or resection specimen at any time within the first 12 months.
Time Frame: 3, 6 and 12 Month
Population: Not all patients in the study were followed for the duration of the treatment phase of 12 months due to study termination. Therefore, primary and secondary endpoint data sample size may vary based on how many visits each subject completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 34
Participants
  3 Month Complete Response | 5
  6 Month Complete Response: number analyzed (Participants) | 30
  6 Month Complete Response | 22
  12 Month Complete Response: number analyzed (Participants) | 16
  12 Month Complete Response | 14

4. Secondary Outcome: Disease Progression Outside the Treatment Area
Description: Proportion of patients demonstrating MGIN or worse outside the TA during treatment phase or follow-up
Time Frame: Initial, 3, 6, 9 and 12 month
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 34
Participants
  Primary RFA | 1
  3-Month: number analyzed (Participants) | 29
  3-Month | 9
  6-Month: number analyzed (Participants) | 16
  6-Month | 6
  9-Month: number analyzed (Participants) | 10
  9-Month | 4
  12-Month: number analyzed (Participants) | 7
  12-Month | 1

ADVERSE EVENTS:
Time Frame: Safety data was evaluated throughout the entirety of follow up, after the study was terminated safety was evaluated for 90 days post RFA procedure.
Arm/Group | Radiofrequency Ablation
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 1/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation (N=34)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
H1N1Influenza (Infections and infestations) | 1 (1)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation (N=34)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early, therefore there was a limited data set for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall not publish the Study results until after Medtronic's multi-site publication or until the elapse of 12 months from the close of the study at all Study sites, whichever occurs earlier.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02953418/SAP_000.pdf
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02953418/Prot_001.pdf